CLINICAL TRIAL: NCT01076647
Title: A 26-week Randomised, Confirmatory, Controlled, Open Label, Multicentre, Multinational Treat-to-target Trial Comparing the Efficacy and Safety of SIBA 200 U/ml Three Times Weekly Injected in the Evening and Insulin Glargine Once Daily in a Population of Insulin naïve Subjects With Type 2 Diabetes Mellitus Currently Treated With OADs Qualifying for Intensified Treatment (BEGIN™: EASY™)
Brief Title: Comparison of NN1250 With Insulin Glargine in Subjects With Type 2 Diabetes
Acronym: BEGIN™
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NN1250-3718; 2009-011399-31 (EudraCT Number); U1111-1112-8770 (Other: WHO)
Record Dates: First submitted 2010-02-25; First posted 2010-02-26 (Estimated); Results first posted 2015-11-10 (Estimated); Last update posted 2017-03-06 (Actual); Status verified 2017-01

CONDITIONS: Diabetes; Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 2 | interventions — insulin degludec; Insulin Glargine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- IDeg 3TW (Experimental)
  Interventions: Drug: insulin degludec
- IGlar OD (Active Comparator)
  Interventions: Drug: insulin glargine

INTERVENTIONS:
Drug: insulin degludec — Will be injected subcutaneously (under the skin) once daily three times weekly.
  Arms: IDeg 3TW
Drug: insulin glargine — Will be injected subcutaneously (under the skin) once daily administered at the same time each day.
  Arms: IGlar OD

SUMMARY:
This trial was conducted in Europe and North America. The aim of this clinical trial was to compare NN1250 (insulin degludec (IDeg)), a soluble insulin basal analogue (SIBA), with insulin glargine (IGlar), as add-on to subject's ongoing treatment with metformin and/or DPP-4 (dipeptyl peptidase 4) inhibitors, in patients with type 2 diabetes being treated with oral anti-diabetic drugs (OADs).

ELIGIBILITY:
Inclusion Criteria:

* Type 2 diabetes (diagnosed clinically) for at least 6 months
* Insulin naïve subjects (allowed are: previous short term insulin treatment up to 14 days; treatment during hospitalisation or during gestational diabetes is allowed for periods longer than 14 days)
* Current treatment: metformin monotherapy or metformin in any combination with insulin secretagogues (sulphonylurea (SU) or glinide), DPP-4 inhibitor, alpha-glucosidase-inhibitor (acarbose) with unchanged dosing for at least 3 months prior to visit 1 with the minimum doses stated: -Metformin: alone or in combination (including fixed combination) 1500 mg daily or maximum tolerated dose (at least 1000 mg daily)-Insulin secretagogue (sulfonylurea (SU) or glinide): minimum half of the daily maximal dose according to local labelling -DPP-4 inhibitor: minimum half of the daily maximal dose according to local labelling -alpha-glucosidase-inhibitor (acarbose): minimum half of the daily maximal dose or maximum tolerated dose
* HbA1c 7.0-10.0 % (both inclusive) by central laboratory analysis
* BMI (Body Mass Index) below or equal to 45.0 kg/m^2

Exclusion Criteria:

* Use within the last 3 months prior to Visit 1 of: Thiazoledinediones (TZDs), Exenatide or Liraglutide
* Cardiovascular disease, within the last 6 months prior to visit 1, defined as: stroke; decompensated heart failure New York Heart Association (NYHA) class III or IV; myocardial infarction; unstable angina pectoris; or coronary arterial bypass graft or angioplasty
* Uncontrolled treated/untreated severe hypertension (systolic blood pressure at least 180 millimetre (mm) mercury (Hg) and/or diastolic blood pressure at least 100 mmHg)
* Pregnancy, breast-feeding, the intention of becoming pregnant or not using adequate contraceptive measures according to local requirements
* Cancer and medical history of cancer hereof (except basal cell skin cancer or squamous cell skin cancer)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 467 (Actual)
Dates: Start 2010-03; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (100):
- United States (63):
  - Novo Nordisk Investigational Site, Birmingham, Alabama
  - Novo Nordisk Investigational Site, Peoria, Arizona
  - Novo Nordisk Investigational Site, Tucson, Arizona
  - Novo Nordisk Investigational Site, Beverly Hills, California
  - Novo Nordisk Investigational Site, Escondido, California
  - Novo Nordisk Investigational Site, La Jolla, California
  - Novo Nordisk Investigational Site, Los Angeles, California
  - Novo Nordisk Investigational Site, Los Banos, California
  - Novo Nordisk Investigational Site, Monterey, California
  - Novo Nordisk Investigational Site, Palm Springs, California
  - Novo Nordisk Investigational Site, Pasadena, California
  - Novo Nordisk Investigational Site, Redondo Beach, California
  - Novo Nordisk Investigational Site, San Mateo, California
  - Novo Nordisk Investigational Site, Tarzana, California
  - Novo Nordisk Investigational Site, Tustin, California
  - Novo Nordisk Investigational Site, Denver, Colorado
  - Novo Nordisk Investigational Site, Golden, Colorado
  - Novo Nordisk Investigational Site, Boynton Beach, Florida
  - Novo Nordisk Investigational Site, DeLand, Florida
  - Novo Nordisk Investigational Site, Kissimmee, Florida
  - Novo Nordisk Investigational Site, Miami, Florida
  - Novo Nordisk Investigational Site, Orange Park, Florida
  - Novo Nordisk Investigational Site, Plantation, Florida
  - Novo Nordisk Investigational Site, Tampa, Florida
  - Novo Nordisk Investigational Site, West Palm Beach, Florida
  - Novo Nordisk Investigational Site, Conyers, Georgia
  - Novo Nordisk Investigational Site, Dunwoody, Georgia
  - Novo Nordisk Investigational Site, Arlington Heights, Illinois
  - Novo Nordisk Investigational Site, Chicago, Illinois
  - Novo Nordisk Investigational Site, Springfield, Illinois
  - Novo Nordisk Investigational Site, Wichita, Kansas
  - Novo Nordisk Investigational Site, Crestview Hills, Kentucky
  - Novo Nordisk Investigational Site, Madisonville, Kentucky
  - Novo Nordisk Investigational Site, Metairie, Louisiana
  - Novo Nordisk Investigational Site, Glen Burnie, Maryland
  - Novo Nordisk Investigational Site, Reisterstown, Maryland
  - Novo Nordisk Investigational Site, Silver Spring, Maryland
  - Novo Nordisk Investigational Site, Ann Arbor, Michigan
  - Novo Nordisk Investigational Site, Eagan, Minnesota
  - Novo Nordisk Investigational Site, Smithtown, New York
  - Novo Nordisk Investigational Site, Staten Island, New York
  - Novo Nordisk Investigational Site, Asheville, North Carolina
  - Novo Nordisk Investigational Site, Burlington, North Carolina
  - Novo Nordisk Investigational Site, Whiteville, North Carolina
  - Novo Nordisk Investigational Site, Winston-Salem, North Carolina
  - Novo Nordisk Investigational Site, Cincinnati, Ohio
  - Novo Nordisk Investigational Site, Dayton, Ohio
  - Novo Nordisk Investigational Site, Altoona, Pennsylvania
  - Novo Nordisk Investigational Site, Harrisburg, Pennsylvania
  - Novo Nordisk Investigational Site, Langhorne, Pennsylvania
  - Novo Nordisk Investigational Site, East Providence, Rhode Island
  - Novo Nordisk Investigational Site, Newberry, South Carolina
  - Novo Nordisk Investigational Site, Chattanooga, Tennessee
  - Novo Nordisk Investigational Site, Kingsport, Tennessee
  - Novo Nordisk Investigational Site, Arlington, Texas
  - Novo Nordisk Investigational Site, Dallas, Texas
  - Novo Nordisk Investigational Site, Houston, Texas
  - Novo Nordisk Investigational Site, Round Rock, Texas
  - Novo Nordisk Investigational Site, Ogden, Utah
  - Novo Nordisk Investigational Site, Salt Lake City, Utah
  - Novo Nordisk Investigational Site, Chesapeake, Virginia
  - Novo Nordisk Investigational Site, Seattle, Washington
  - Novo Nordisk Investigational Site, Spokane, Washington
- Bulgaria (4):
  - Novo Nordisk Investigational Site, Burgas
  - Novo Nordisk Investigational Site, Rousse
  - Novo Nordisk Investigational Site, Sofia
  - Novo Nordisk Investigational Site, Stara Zagora
- Canada (5):
  - Novo Nordisk Investigational Site, Chilliwack, British Columbia
  - Novo Nordisk Investigational Site, Ottawa, Ontario
  - Novo Nordisk Investigational Site, Thornhill, Ontario
  - Novo Nordisk Investigational Site, Toronto, Ontario
  - Novo Nordisk Investigational Site, Québec, Quebec
- France (8):
  - Novo Nordisk Investigational Site, La Roche-sur-Yon
  - Novo Nordisk Investigational Site, La Rochelle
  - Novo Nordisk Investigational Site, Le Creusot
  - Novo Nordisk Investigational Site, Nanterre
  - Novo Nordisk Investigational Site, Narbonne
  - Novo Nordisk Investigational Site, Nîmes
  - Novo Nordisk Investigational Site, Paris
  - Novo Nordisk Investigational Site, Vénissieux
- Hungary (6):
  - Novo Nordisk Investigational Site, Budapest
  - Novo Nordisk Investigational Site, Debrecen
  - Novo Nordisk Investigational Site, Eger
  - Novo Nordisk Investigational Site, Gyula
  - Novo Nordisk Investigational Site, Kaposvár
  - Novo Nordisk Investigational Site, Szeged
- Netherlands (8):
  - Novo Nordisk Investigational Site, Amsterdam
  - Novo Nordisk Investigational Site, Beek
  - Novo Nordisk Investigational Site, Etten-Leur
  - Novo Nordisk Investigational Site, Hengelo
  - Novo Nordisk Investigational Site, Hoogeveen
  - Novo Nordisk Investigational Site, Lieshout
  - Novo Nordisk Investigational Site, Utrecht
  - Novo Nordisk Investigational Site, Zwijndrecht
- Romania (6):
  - Novo Nordisk Investigational Site, Oradea, Bihor County
  - Novo Nordisk Investigational Site, Satu Mare, Satu Mare County
  - Novo Nordisk Investigational Site, Bacau
  - Novo Nordisk Investigational Site, Botoșani
  - Novo Nordisk Investigational Site, Bucharest
  - Novo Nordisk Investigational Site, Galati

REFERENCES:
- [Result] Zinman B, DeVries JH, Bode B, Russell-Jones D, Leiter LA, Moses A, Johansen T, Ratner R; NN1250-3724 (BEGIN:EASY AM) and NN1250-3718 (BEGIN:EASY PM) Trial Investigators. Efficacy and safety of insulin degludec three times a week versus insulin glargine once a day in insulin-naive patients with type 2 diabetes: results of two phase 3, 26 week, randomised, open-label, treat-to-target, non-inferiority trials. Lancet Diabetes Endocrinol. 2013 Oct;1(2):123-31. doi: 10.1016/S2213-8587(13)70013-5. Epub 2013 Jul 9. PMID 24622318
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The trial was conducted at 89 sites in 7 countries: Bulgaria, Canada, France, Hungary, Netherlands, Romania, and United States.
Groups:
- IDeg 3TW: Insulin degludec (IDeg) 200 U/ml was given thrice weekly on Mondays, Wednesdays and Fridays subcutaneously (s.c.) in the evening with pre-trial metformin and with or without pre-trial DPP-4 for 26 weeks.
- IGlar OD: Insulin glargine (IGlar) was given once daily (OD) subcutaneously (s.c.) same time each day according to local labelling with pre-trial metformin and with or without pre-trial DPP-4 for 26 weeks.
Period: Overall Study
Arm/Group | IDeg 3TW | IGlar OD
Started | 233 | 234
Completed | 208 | 209
Not Completed | 25 | 25
Not completed — Adverse Event | 4 | 1
Not completed — Lack of Efficacy | 0 | 1
Not completed — Protocol Violation | 7 | 9
Not completed — Withdrawal criteria | 2 | 2
Not completed — Unclassified | 12 | 12

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | IDeg 3TW | IGlar OD | Total
Number analyzed (Participants) | 233 | 234 | 467
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.3 (9.6) | 57.5 (10.7) | 57.4 (10.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 101 | 99 | 200
  Male | 132 | 135 | 267
Glycosylated haemoglobin (HbaA1c) [Mean (Standard Deviation); unit: percentage of glycosylated haemoglobin] | 8.3 (0.8) | 8.3 (0.8) | 8.3 (0.8)
Body Weight [Mean (Standard Deviation); unit: kg] | 92.3 (18.3) | 91.4 (18.7) | 91.8 (18.5)

OUTCOME MEASURES:

1. Primary Outcome: Change in Glycosylated Haemoglobin (HbA1c)
Description: Change from baseline in HbA1c after 26 weeks of treatment
Time Frame: Week 0, Week 26
Population: The Full analysis set (FAS) included all randomised subjects and missing data is imputed using last observation carried forward (LOCF).
Measure: Mean (Standard Deviation); unit: percentage of glycosylated haemoglobin
Arm/Group | IDeg 3TW | IGlar OD
Number analyzed (Participants) | 233 | 234
percentage of glycosylated haemoglobin | -1.05 (0.94) | -1.36 (0.95)

2. Secondary Outcome: Change in Body Weight
Description: Change from baseline in body weight after 26 weeks of treatment
Time Frame: Week 0, Week 26
Population: The FAS included all randomised subjects and missing data is imputed using last observation carried forward (LOCF).
Measure: Mean (Standard Deviation); unit: kg
Arm/Group | IDeg 3TW | IGlar OD
Number analyzed (Participants) | 233 | 234
kg | 0.8 (3.9) | 0.5 (3.7)

ADVERSE EVENTS:
Time Frame: The adverse events were collected in a time frame of 26 weeks + 7 days follow up
Description: Safety analysis set includes all subjects who received at least one dose of the investigational product or its comparator.
Arm/Group | IDeg 3TW | IGlar OD
Serious Adverse Events (participants affected / at risk) | 13/233 | 12/234
Other Adverse Events (participants affected / at risk) | 34/233 | 25/234
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | IDeg 3TW (N=233) | IGlar OD (N=234)
Lymphadenopathy (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Angina pectoris (Cardiac disorders) | 0 (0) | 1 (1)
Angina unstable (Cardiac disorders) | 1 (1) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 1 (1)
Cardiac asthma (Cardiac disorders) | 0 (0) | 1 (1)
Tachycardia (Cardiac disorders) | 1 (1) | 0 (0)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Periodontitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Chest pain (General disorders) | 0 (0) | 1 (1)
Erysipelas (Infections and infestations) | 0 (0) | 2 (2)
Road traffic accident (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Hypoglycaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hyponatraemic syndrome (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Intervertebral disc disorder (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Facial paresis (Nervous system disorders) | 0 (0) | 1 (1)
Presyncope (Nervous system disorders) | 0 (0) | 1 (1)
Vertebrobasilar insufficiency (Nervous system disorders) | 0 (0) | 1 (1)
Vertigo CNS origin (Nervous system disorders) | 1 (1) | 0 (0)
Depression (Psychiatric disorders) | 0 (0) | 1 (1)
Panic disorder (Psychiatric disorders) | 0 (0) | 1 (1)
Ovarian cyst (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Lithotripsy (Surgical and medical procedures) | 1 (1) | 0 (0)
Arteriosclerosis (Vascular disorders) | 0 (0) | 1 (1)
Deep vein thrombosis (Vascular disorders) | 1 (1) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | IDeg 3TW (N=233) | IGlar OD (N=234)
Diarrhoea (Gastrointestinal disorders) | 11 (13) | 13 (16)
Nasopharyngitis (Infections and infestations) | 13 (14) | 6 (6)
Headache (Nervous system disorders) | 14 (18) | 8 (9)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Novo Nordisk maintains the right to be informed of any Investigator plans for publication and to review any scientific paper, presentation, communication or other information concerning the investigation described in this protocol. Any such communication must be submitted in writing to the Novo Nordisk trial manager prior to submission for comments. Comments will be given within four weeks from receipt of the planned communication.